CLINICAL TRIAL: NCT05573048
Title: Optical Fusion Trans-Perineal Grid
Brief Title: A Study of Optical Fusion Trans-Perineal Grid
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Clear Guide Medical Inc. (Unknown)
Responsible Party: Principal Investigator, David A. Woodrum, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 22-003369
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Prostate Biopsy
Keywords: Prostate Ablation Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Trans-Perineal Grid for prostate interventions (Experimental): Subjects will have the trans-perineal guide grid placed the prostate biopsy or ablation procedure.
  Interventions: Device: Trans-Perineal Grid

INTERVENTIONS:
Device: Trans-Perineal Grid — A small square piece of plastic with many holes in it placed between the legs to help guide the path of the interventional instruments and to facilitate the prostate intervention. The guide grid will help with needle placement using the grid technology.

SUMMARY:
The purpose of this research is to evaluate a new needle guide grid utilizing Clear Guide SCENERGY - MR with a grid embedded with VisiMARKER II to autoregister and target the prostate aiding in needle placement positioning. The proceduralist can utilize this technology to find the best needle path to target within the pelvis.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a MR guided biopsy or ablation.
* One, two, or three tumor suspicious regions identified on multiparametric MRI.
* Tolerance for anesthesia/sedation.
* Ability to give informed consent.

Exclusion Criteria:

* Presence of any condition (e.g., metal implant, shrapnel) not compatible with MRI.
* History of other primary non-skin malignancy within previous three years.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Needle placement accuracy | Baseline
  Number of needle placements to successfully match target and needle tip position assessed by direct MR imaging and

CONTACTS AND LOCATIONS:
Overall Officials: David Woodrum, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials